CLINICAL TRIAL: NCT06117358
Title: Detection of Pre-Diabetes in Overweight and Obese Children and Adolescents in Assiut Governorate
Brief Title: Detection of Pre-Diabetes in Overweight and Obese Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Bakr Gaber, Principal Investigator, Assiut University
Other Study IDs: Detection of Pre-Diabetes
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pre-Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — Descriptive cross section study

SUMMARY:
Descriptive cross section study To detect prediabetes in overweight and obese children and adolescents in Assiut Governorate and to find out the possible risk factors.

DETAILED DESCRIPTION:
Childhood obesity has reached epidemic levels in developed as well as in developing countries, Overweight and obesity in childhood have significant impact on both physical and psychological health.

Childhood obesity has been linked to numerous medical conditions. These conditions include : fatty liver disease, sleep apnea, Type 2 diabetes, asthma, cardiovascular disease, high cholesterol, cholelithiasis (gallstones), glucose intolerance and insulin resistance, etc.

Obesity is associated with Prediabetes , a significant risk factor for development of type 2 diabetes mellitus T2DM and its accompanying complications.

In some populations, type 2 diabetes is now the dominant form of diabetes in children and adolescents.

Prediabetes is defined by a fasting glucose level of 100 to 125 mg/dL , glycated hemoglobin level (HbA1C) of 5.7% to 6.4% , or a glucose level of 140 to 199 mg/dL measured 2 hours after a 75-g oral glucose load. approximately 10% of people with prediabetes progress to having diabetes each year.

The vast majority of pediatric cases occur after age 10, with the peak age for presentation occurring at mid-puberty (approximately age 14 years).

The ADA recommends screening for type 2 diabetes in children after onset of puberty or age 10 years who are overweight (BMI ≥85th percentile) or obese (BMI ≥95th percentile) and have one or more additional risk factors for diabetes.

One report in JAMA Pediatrics found that nearly one in three adolescents and teens has prediabetes and the rate among 12 to 19 year-olds more than doubled between 1999-2002 and 2015-2018, jumping from 12 percent to 28 percent.

However , no enough data are available regarding prevalence and risk factors of prediabetes in overweight and obese youth particularly in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes , aged (10-18) years.
* Body mass index calculated as weight in Kg/(height in meters)2 :

  * Over weight > 85% percentile
  * Obese > 95% percentile " On Egyptian growth chart "

Exclusion Criteria:

* • Children and adolescents with type 2 diabetes mellitus.

  * Children and adolescents with drug history affecting blood glucose level as corticosteroids.
  * Children and adolescents with any condition affecting blood glucose level as Cushing disease.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: • obese and overweight children and adolescents in Assiut governorate aged between (10-18) years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Pre-Diabetes in Overweight and Obese children and adolescents in Assiut governorate | Baseline
  determine the prevalence of prediabetes in overweight and obese children and adolescents in Assiut Governorate and to find out the possible risk factors through many investigations as HbA1c , Fasting blood glucose level , Lipid profile in 150 obese children.